CLINICAL TRIAL: NCT05235126
Title: A Post-market, Prospective, Observational (Non-interventional), Partly Confirmatory, Multi-centre Clinical Investigation to Confirm the Clinical Safety and Performance Profile of Decoria® Intense Hyaluronic Acid Dermal Filler for the Correction of Nasolabial Folds.
Brief Title: A Clinical Investigation of the Decoria® Aesthetic Group (DAG) for Correction of Nasolabial Folds (NLF)
Acronym: Decorate01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bohus Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Decorate01
Record Dates: First submitted 2022-01-27; First posted 2022-02-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-07

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: All subjects will receive open treatment with Decoria intense for correction of nasolabial folds at Visit 1 with optional touch-up at Visit 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Other): All subjects receive treatment at V1 and option to receive touch-up at V2.
  Interventions: Device: Decoria intense

INTERVENTIONS:
Device: Decoria intense — All subjects will receive treatment at Visit 1 with the option to receive a touch-up treatment at Visit 2. Evaluation of the nasolabial folds will be performed by PI using the Wrinkle Severity Rating Scale (WSRS).

SUMMARY:
Decoria intense is a class III medical device and is CE-marked and has been on the market since 2014. Decoria intense is a hyaluronic acid filler that will be used according to intended use for correction of nasolabial folds.

According to the new MDR in EU this clinical investigation will confirm efficacy and safety of Decoria intense.

The plan is to recruit 80 subjects to receive 64 evaluable subjects during 6 months recruitment.

The clinical investigation contains 5 visits and the total time per subject is 12 months. All subjects will receive treatment at Visit 1 with the option to receive a touch-up treatment at Visit 2. Evaluation of the nasolabial folds will be performed by PI using the Wrinkle Severity Rating Scale (WSRS)

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, ≥18 years of age, of all weight spans, desiring correction of their nasolabial folds.
2. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the Informed Consent Form (ICF).
3. The subject has nasolabial folds considered at least moderate (grade 3) according to the Wrinkle Severity Rating Scale (WSRS), as assessed by the Principal Investigator.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any previous hypersensitivity reaction to any constituent of the Investigational medical device (IMD) or to local anaesthetic products.
3. Any acute or chronic skin disease or inflammation (such as pimples, rashes or hives) within or close to the area selected for correction.
4. Any bleeding disorder or treatment with thrombolytics or anticoagulants.
5. Any treatment with interferon and ribavirin.
6. Any vaccine taken within 2 weeks prior to the treatment visit.
7. Any other intradermal injection, such as fillers or toxins, received in the same injection area within 6 months of the Screening and Treatment visit (Visit 1).
8. Participation in a clinical investigation study that may affect the safety or performance of this investigation, within one year of enrolment, or planned participation in such investigation at any time during this clinical investigation, as judged by the Principal Investigator.
9. Any other condition or treatment making the subject unsuitable for participation in the clinical investigation, as judged by the Principal Investigator.
10. Employees of the study site or the sponsor directly involved with the conduct of the investigation, or immediate family members of any such individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Change in the WSRS score | 3 months after pre-treatment (baseline)
  The primary efficacy endpoint is to measure the change in the WSRS score from pre-treatment baseline, at 3 months post OCR, as assessed by the Principal Investigator. The WSRS range from 1 (absent - no visible fold) to 5 (extreme - extremely deep and long folds). A subject improving 1 score or more is classified as "responder". A stable subject or a subject worsening is classified as "non-responder".
The rate of adverse events | 12 months.
  The primary safety endpoint is to assess the safety of Decoria® intense, evaluated by the rate of adverse events throughout the study period.

SECONDARY OUTCOMES:
Subject satisfaction with treatment | 12 months
  The subject will assess the satisfaction with the treatment at all visits using the Global Aesthetic Improvement Scale (GAIS) 1 - 5. 1. Exceptional improvement, 2. Very improved patient, 3. Improved patient, 4. Unaltered patient, 5. Worsened patient.
PI satisfaction with treatment | 6 months
  The PI will assess the satisfaction with the treatment at all visits except for visit 5 (telephone visit) using the Global Aesthetic Improvement Scale (GAIS) 1 - 5. 1. Exceptional improvement, 2. Very improved patient, 3. Improved patient, 4. Unaltered patient, 5. Worsened patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Grema, MD, Principal Investigator — Florakliniken Stockholm Sweden
Locations (2):
- Sweden (2):
  - MyBeauty Clinic, Halmstad
  - Florakliniken, Stockholm

IPD SHARING:
Plan to Share IPD: No